CLINICAL TRIAL: NCT05743062
Title: Awe Inducing Elements in Virtual Reality Applications: A Prospective Study of Hospitalized Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 69170
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Awe
Keywords: Virtual Reality

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Virtual reality intervention will be given 6 times in total and each session will last not more than 60 seconds.
  Interventions: Behavioral: Virtual Reality
- Control (Other): Participants will serve as their own controls. Participants will not be given any VR intervention at first but they are requested to fill out the survey to collect the baseline data.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Virtual Reality — Virtual reality intervention will be given 6 times in total and each session will last not more than 60 seconds. Participants will be asked to fill out a survey before the intervention to collect the baseline data, after each session of VR intervention and a final survey at the end of the study.
  Arms: Virtual Reality
Other: Control — For case control, participants will service as their self control and no VR intervention will be given at first. Participants will be asked to fill out a survey before the intervention to collect the baseline data.
  Arms: Control

SUMMARY:
This is an experimental study to evaluate which aspects of virtual reality (VR) software development can be optimized to increase awe in pediatric perioperative patients and their adult caregivers (e.g., parents, guardians)

DETAILED DESCRIPTION:
Hospitalized pediatric patients, especially those undergoing anesthesia and surgery, experience anxiety and fear, resulting in lack of cooperation, withdrawal, and aggression. These reactions delay medical care and negatively impact patient experience.

This is an experimental, prospective study to evaluate which aspects of virtual reality (VR) software development can be optimized to increase awe in pediatric perioperative patients and their adult caregivers. The primary center for this study will be Lucile Packard Children's Hospital Stanford (LPCHS) (located within Stanford University, Palo Alto, CA).

After software development, we will evaluate the awe and engagement of pediatric patients after experiencing the novel virtual reality application.

ELIGIBILITY:
Inclusion Criteria:

* Patient with age range from 6 to 25
* Adult or LAR with age range from 18 to 99
* Able to consent or have parental consent
* in pre-operative holding and inpatient acute care areas of LCPH
* English speaking participants

Exclusion Criteria:

* People who do not consent
* Significant Cognitive Impairment
* History of Severe Motion Sickness
* Visual Problems
* currently have nausea
* history of seizures
* non-english participants

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Change in awe levels measured by Global Perceived Awe Survey | Duration of intervention, approximately 20-30 minutes
  Global Perceived Awe Survey contains an 7-point Likert scale . Scores range from 1 (strongly disagree) to 7 (Strongly agree), with higher score indicates strongly agree to the statement.

SECONDARY OUTCOMES:
Change in engagement measured by Game Engagement Questionnaire | Duration of intervention, approximately 20-30 minutes
  Game Engagement Questionnaire contains 19 items . Scores range from 1 (strongly disagree) to 7 (Strongly agree), with higher score indicates strongly agree to the statement.
Change in awe levels measured by Perceived Vastness Survey | Duration of intervention, approximately 20-30 minutes
  Perceived Vastness Survey contains 4 items . Scores range from 1 (strongly disagree) to 7 (Strongly agree), with higher score indicates strongly agree to the statement.
Change in awe levels measured by Perceived Need for Accommodation Survey | Duration of intervention, approximately 20-30 minutes
  Perceived Need for Accommodation Survey contains 3 items . Scores range from 1 (strongly disagree) to 7 (Strongly agree), with higher score indicates strongly agree to the statement.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Parkard Children's Hospital, Stanford, California, United States

REFERENCES:
- [Background] Chirico A, Cipresso P, Yaden DB, Biassoni F, Riva G, Gaggioli A. Effectiveness of Immersive Videos in Inducing Awe: An Experimental Study. Sci Rep. 2017 Apr 27;7(1):1218. doi: 10.1038/s41598-017-01242-0. PMID 28450730
- [Background] Rodriguez CM, Clough V, Gowda AS, Tucker MC. Multimethod assessment of children's distress during noninvasive outpatient medical procedures: child and parent attitudes and factors. J Pediatr Psychol. 2012 Jun;37(5):557-66. doi: 10.1093/jpepsy/jss005. Epub 2012 Mar 16. PMID 22427698
- [Background] Chon T, Ma A, Mun-Price C. Perioperative Fasting and the Patient Experience. Cureus. 2017 May 24;9(5):e1272. doi: 10.7759/cureus.1272. PMID 28652955
- [Background] Chirico A, Ferrise F, Cordella L, Gaggioli A. Designing Awe in Virtual Reality: An Experimental Study. Front Psychol. 2018 Jan 22;8:2351. doi: 10.3389/fpsyg.2017.02351. eCollection 2017. PMID 29403409
- [Background] Caruso TJ, O'Connell C, Qian JJ, Kung T, Wang E, Kinnebrew S, Pearson M, Kist M, Menendez M, Rodriguez ST. Retrospective Review of the Safety and Efficacy of Virtual Reality in a Pediatric Hospital. Pediatr Qual Saf. 2020 Apr 10;5(2):e293. doi: 10.1097/pq9.0000000000000293. eCollection 2020 Mar-Apr. PMID 32426648
- [Background] Richey AE, Hastings KG, Karius A, Segovia NA, Caruso TJ, Frick S, Rodriguez S. Virtual Reality Reduces Fear and Anxiety During Pediatric Orthopaedic Cast Room Procedures: A Randomized Controlled Trial. J Pediatr Orthop. 2022 Nov-Dec 01;42(10):600-607. doi: 10.1097/BPO.0000000000002250. Epub 2022 Aug 30. PMID 36040069
- [Background] Tas FQ, van Eijk CAM, Staals LM, Legerstee JS, Dierckx B. Virtual reality in pediatrics, effects on pain and anxiety: A systematic review and meta-analysis update. Paediatr Anaesth. 2022 Dec;32(12):1292-1304. doi: 10.1111/pan.14546. Epub 2022 Sep 1. PMID 35993398
- [Background] Eijlers R, Utens EMWJ, Staals LM, de Nijs PFA, Berghmans JM, Wijnen RMH, Hillegers MHJ, Dierckx B, Legerstee JS. Systematic Review and Meta-analysis of Virtual Reality in Pediatrics: Effects on Pain and Anxiety. Anesth Analg. 2019 Nov;129(5):1344-1353. doi: 10.1213/ANE.0000000000004165. PMID 31136330
- [Background] Gao Y, Xu Y, Liu N, Fan L. Effectiveness of virtual reality intervention on reducing the pain, anxiety and fear of needle-related procedures in paediatric patients: A systematic review and meta-analysis. J Adv Nurs. 2023 Jan;79(1):15-30. doi: 10.1111/jan.15473. Epub 2022 Nov 3. PMID 36330583
- See also: The development of the Game Engagement Questionnaire: A measure of engagement in video game-playing. — https://www.semanticscholar.org/paper/EFFECT-OF-OPERATIVE-PROCEDURES-ON-THE-EMOTIONAL-OF-Pearson/3cd20d7f33c26882edb7a4df4650b81f495702a3
- See also: The development of the Awe Experience Scale (AWE-S): A multifactorial measure for a complex emotion — https://scottbarrykaufman.com/wp-content/uploads/2018/07/The-development-of-the-Awe-Experience-Scale-AWE-S-A-multifactorial-measure-for-a-complex-emotion.pdf